CLINICAL TRIAL: NCT01755234
Title: The Effects of Propofol vs. Sevoflurane Administered During Anesthesia Maintenance on Early and Late Recovery After Gynecological Surgery
Brief Title: Propofol Versus Sevoflurane Recovery After Gynecological Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Prinipal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00070833
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Surgery; Anesthesia
Keywords: Outpatient; Surgery; Anesthesia
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): Sevoflurane administered by inhalation (laryngeal mask airway or endotracheal tube)
  Interventions: Drug: Sevoflurane
- Propofol (Active Comparator): Propofol administered via intravenous catheter at an initial rate of 1.0 -2.0 mg/kg then the Propofol infusion rate will be titrated to keep a bispectral index between 40-60
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevfoflurane inhaled administered by laryngeal mask airway or endotracheal tube
  Other Names: Sevoflurane,Ultane
  Arms: Sevoflurane
Drug: Propofol — Propofol administered via intravenous catheter at an initial rate of 1.0 -2.0 mg/kg then the Propofol infusion rate will be titrated to keep a bispectral index between 40-60
  Other Names: Propofol,Diprivan
  Arms: Propofol

SUMMARY:
80% of 25 million American who undergo surgery describe moderate to severe pain. The use of multimodal analgesic techniques can attenuate patient's postoperative pain and several different medication have been found to be effective. Pain can significantly affect patient's quality of recovery after surgery. Volatile anesthetics can increase sensitivity to pain at the low concentrations present on emergence from anesthesia. Propofol may have analgesic effect at sedative doses. The effects of propofol,when used for anesthesia maintenance, on postoperative pain have demonstrated controversial results with some investigators showing a potential benefit whereas others have not shown any benefit. Propofol for maintenance of anesthesia has been advocated as an strategy for high risk patients even though it has shown controversial results on reduction of Post operative nausea and vomiting. A comparison of propofol vs.volatile anesthetic in regards to the time required by patients to meet discharge criteria has also shown conflicting results.The QOR 40 is a validated instrument that has been specifically developed to evaluate patients recovery after anesthesia and surgery.

The purpose of this study is to compare the effects of maintenance of anesthesia with two agents (Propofol and Sevoflurane) on quality of recovery after ambulatory surgery

Significance: the results of this study can lead to the discovery of an anesthesia technique that is associated with a better recovery for patients after ambulatory surgery.

Research question is: do patients anesthetized with propofol have a better quality of recovery after ambulatory anesthesia than patients anesthetized with Sevoflurane? The hypothesis: patients anesthetized with propofol will have better quality of recovery than patients anesthetized with Sevoflurane after ambulatory surgery.

DETAILED DESCRIPTION:
Subjects will be recruited up to the day of surgery. 90 subjects will be randomly allocated into 2 groups, using a computer generated table of random numbers: anesthetic maintenance with Sevoflurane or anesthetic maintenance with Propofol . Subjects will be premedicated with intravenous (IV) midazolam 0.04 mg/kg. Routine ASA monitors will be applied. Anesthesia will be induced with remifentanil infusion started at 0.1 mcg/kg/minute titrated to keep blood pressure within 20% of the baseline and propofol 1.0 -2.0 mg/kg or sevoflurane induction. Tracheal intubation will be facilitated with rocuronium (0.6 mg/kg) or succinylcholine (1-2mg /kg). Anesthesia will be maintained with Sevoflurane or a Propofol infusion titrated to keep a bispectral index between 40-60, remifentanil infusion started at 0.1mcg/kg/min titrated to keep blood pressure within 20 % of baseline values, and rocuronium that will be administered at the discretion of the anesthesiologist. Upon termination of the surgery, neuromuscular blockade will be antagonized with a combination of neostigmine 0.05mg/kg and glycopyrrolate 0.01 mg/kg. Subjects will also receive Ketorolac 30 mg IV after discontinuation of remifentanil for postoperative pain control. Ondansetron 4 mg IV will be administered to decrease postoperative nausea and vomiting. Subjects will receive IV hydromorphone 0.4 mg q 5 minutes as needed to achieve a verbal rating score for pain <4 out of 10.They will also receive reglan 10 mg IV as a rescue antiemetic, if not effective, a second dose of Zofran 4 mg IV will be given in PACU. 24 hours after surgery a QOR 40 will be administered to the patient by one of the investigators. The primary and secondary outcomes will be assessed by an independent observer who will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-64
* Patients undergoing ambulatory surgery
* ASA PS I, II

Exclusion Criteria:

* Chronic opioid use
* Pregnant patient

Drop Out : patient or surgeon request

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White PF, Kehlet H. Improving postoperative pain management: what are the unresolved issues? Anesthesiology. 2010 Jan;112(1):220-5. doi: 10.1097/ALN.0b013e3181c6316e. No abstract available. PMID 20010418
- [Background] White PF. The changing role of non-opioid analgesic techniques in the management of postoperative pain. Anesth Analg. 2005 Nov;101(5 Suppl):S5-S22. doi: 10.1213/01.ANE.0000177099.28914.A7. PMID 16334489
- [Background] Zhang Y, Eger EI 2nd, Dutton RC, Sonner JM. Inhaled anesthetics have hyperalgesic effects at 0.1 minimum alveolar anesthetic concentration. Anesth Analg. 2000 Aug;91(2):462-6. doi: 10.1097/00000539-200008000-00044. PMID 10910869
- [Background] Hand R Jr, Riley GP, Nick ML, Shott S, Faut-Callahan M. The analgesic effects of subhypnotic doses of propofol in human volunteers with experimentally induced tourniquet pain. AANA J. 2001 Dec;69(6):466-70. PMID 11837149
- [Background] Cheng SS, Yeh J, Flood P. Anesthesia matters: patients anesthetized with propofol have less postoperative pain than those anesthetized with isoflurane. Anesth Analg. 2008 Jan;106(1):264-9, table of contents. doi: 10.1213/01.ane.0000287653.77372.d9. PMID 18165589
- [Background] Boccara G, Mann C, Pouzeratte Y, Bellavoir A, Rouvier A, Colson P. Improved postoperative analgesia with isoflurane than with propofol anaesthesia. Can J Anaesth. 1998 Sep;45(9):839-42. doi: 10.1007/BF03012216. PMID 9818105
- [Background] Visser K, Hassink EA, Bonsel GJ, Moen J, Kalkman CJ. Randomized controlled trial of total intravenous anesthesia with propofol versus inhalation anesthesia with isoflurane-nitrous oxide: postoperative nausea with vomiting and economic analysis. Anesthesiology. 2001 Sep;95(3):616-26. doi: 10.1097/00000542-200109000-00012. PMID 11575532
- [Background] Watson KR, Shah MV. Clinical comparison of 'single agent' anaesthesia with sevoflurane versus target controlled infusion of propofol. Br J Anaesth. 2000 Oct;85(4):541-6. doi: 10.1093/bja/85.4.541. PMID 11064611
- [Background] Rohm KD, Piper SN, Suttner S, Schuler S, Boldt J. Early recovery, cognitive function and costs of a desflurane inhalational vs. a total intravenous anaesthesia regimen in long-term surgery. Acta Anaesthesiol Scand. 2006 Jan;50(1):14-8. doi: 10.1111/j.1399-6576.2006.00905.x. PMID 16451145 (Retraction: PMID 21749337 Acta Anaesthesiol Scand. 2011 Aug;55(7):903)
- [Background] Montes FR, Trillos JE, Rincon IE, Giraldo JC, Rincon JD, Vanegas MV, Charris H. Comparison of total intravenous anesthesia and sevoflurane-fentanyl anesthesia for outpatient otorhinolaryngeal surgery. J Clin Anesth. 2002 Aug;14(5):324-8. doi: 10.1016/s0952-8180(02)00367-7. PMID 12208434
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Derived] De Oliveira GS Jr, Bialek J, Rodes ME, Kendall MC, McCarthy RJ. The effect of sevoflurane compared to propofol maintenance on post-surgical quality of recovery in patients undergoing an ambulatory gynecological surgery: A prospective, randomized, double-blinded, controlled, clinical trial. J Clin Anesth. 2017 Dec;43:70-74. doi: 10.1016/j.jclinane.2017.10.001. Epub 2017 Oct 13. PMID 29032007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited 12/2012-04/2014. 101 subjects were assessed for eligibility, 4 did not meet inclusion criteria and 7 declined to participate. 90 subjects were randomized.
Period: Overall Study
Arm/Group | Sevoflurane | Propofol
Started | 45 | 45
Completed | 30 | 37
Not Completed | 15 | 8
Not completed — Lost to Follow-up | 11 | 6
Not completed — Change in surgical case | 2 | 1
Not completed — case cancelled | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — unblinded | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane | Propofol | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Score 24 Hours Post Operative
Description: Quality of recovery score 24 hours after the surgical procedure.Score of 40 is poor recovery and a score of 200 is good recovery.
Time Frame: 24 hours after the surgical procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Sevoflurane | Propofol
Number analyzed (Participants) | 30 | 37
units on a scale | 175 [163 to 181] | 176 [163 to 184]
Statistical Analysis 1: Comparison: Sevoflurane vs Propofol; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Mg of Morphine Equivalents (IV)
Description: Total opioid use in the post operative care unit (Mg of morphine equivalents)
Time Frame: PACU admission to discharge
Measure: Median (Inter-Quartile Range); unit: miligrams of morphine equivalents
Arm/Group | Sevoflurane | Propofol
Number analyzed (Participants) | 30 | 37
miligrams of morphine equivalents | 9 [4 to 17] | 9.4 [5 to 17]
Statistical Analysis 1: Comparison: Sevoflurane vs Propofol; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain in Post Anesthesia Care Unit
Description: Numeric rating scale for pain on a scale of 0-10 (0 is no pain and 10 is high pain) versus time curve in the post anesthesia care unit ( score * min). A higher value indicates more pain and time in the Post Anesthesia Care Unit.
  The range is 0 pain to x time in minutes x 1 hour to 5 hour ( 60-300 minutes) . The pain scores were collected at 15 minute intervals from the time of admission to the PACU. The area under the NRS pain scale versus time curve was calculated using the trapezoidal method as an indicator of pain burden during early recovery (Graph Pad Prism ver 5.03, Graph Pad Software INC.
Time Frame: Time in the post anesthesia care unit
Measure: Median (Inter-Quartile Range); unit: Pain Score * minutes in PACU
Arm/Group | Sevoflurane | Propofol
Number analyzed (Participants) | 30 | 37
Pain Score * minutes in PACU | 270 [195 to 330] | 240 [165 to 330]
Statistical Analysis 1: Comparison: Sevoflurane vs Propofol; Test type: Superiority or Other; p = .96, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Opioid Use Discharge From Post Anesthesia Care Unit to 24 Hours After PACU Discharge.
Description: Opioid use in mg of morphine equivalents from discharge from the post anesthesia care unit to 24 hours after PACU discharge.
Time Frame: Discharge from PACU to 24 hours post operative after PACU discharge.
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Sevoflurane | Propofol
Number analyzed (Participants) | 30 | 37
mg morphine equivalents | 30 [10 to 40] | 25 [0 to 40]
Statistical Analysis 1: Comparison: Sevoflurane vs Propofol; Test type: Superiority or Other; p = .84, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Time in the post anesthesia care unit.
Description: Nausea experienced in the post anesthesia care unit
Arm/Group | Sevoflurane | Propofol
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/37
Other Adverse Events (participants affected / at risk) | 13/30 | 11/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevoflurane (N=30) | Propofol (N=37)
Nausea (Gastrointestinal disorders) | 13 (13) | 11 (11) — Development of nausea during the post operative period in the post operative care unit.
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) — Vomiting during the post operative period in the post anesthesia care unit.

LIMITATIONS AND CAVEATS:
We only studied patients undergoing outpatient laparoscopic gynecological surgery, therefore, our results cannot be generalizable to other surgical procedures.

We also administered remifentanil which is has been linked to hyperalgesia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes